CLINICAL TRIAL: NCT01694901
Title: Optimization of the Anesthetic Regimen Using the SmartPilot® System and Influence on Different Outcome Parameters - a Pilot Study. A Single- Center Prospective Randomized Controlled Pilot Study.
Brief Title: Optimization of the Anesthetic Regimen Using the SmartPilot® System and Influence on Different Outcome Parameters - a Pilot Study.
Status: Completed | Type: Observational
Sponsor: Claudia Spies (Other)
Responsible Party: Sponsor-Investigator, Claudia Spies, Prof. Dr. C. Claudia, Charite University, Berlin, Germany
Organization: Charite University, Berlin, Germany (Other)
Other Study IDs: Smart-Outcome
Record Dates: First submitted 2012-09-25; First posted 2012-09-27 (Estimated); Last update posted 2019-06-28 (Actual); Status verified 2019-06

CONDITIONS: Postoperative Cognitive Disturbances

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- SmartPilot® system: 50 patients scheduled for elective surgery (general/abdominal surgery; traumatological/orthopedic surgery, gynecology, urology) in general anesthesia using the SmartPilot® system
- Standard arm: 50 patients scheduled for elective surgery (general/abdominal surgery; traumatological/orthopedic surgery, gynecology, urology) in general anesthesia according to the standard operating procedures of the department, i.e. manually controlled clinical anesthesia and EEG-derived parameters of anesthetic depth

SUMMARY:
This study investigates whether general anesthesia using a Pharmacokinetic/Pharmacodynamic (PK/PD) -model-based index indicating the compound effect of different anesthetics leads to optimized outcome compared to manually controlled clinical anesthesia and computerized Electroencephalogram (EEG).

ELIGIBILITY:
Inclusion Criteria:

* Offered patient information and written informed consent
* Male/female patients with intended ratio of 1:1
* patients aged greater than or equal to 60 years
* scheduled duration of surgery longer than or equal to 60 minutes
* elective surgery (general/abdominal surgery, traumatological/orthopedic surgery, gynecology, urology) in general anesthesia

Exclusion Criteria:

* Persons without the capacity to consent
* Unability of German language use
* Lacking willingness to save and hand out data within the study
* Participation in another study according to the German Medicinal Products Act within 30 days before participation in the Smart-Outcome study
* Accommodation in an institution due to an official or judicial order
* (Unclear) history of alcohol or substances disabuse
* Member of staff of the Charité
* Neurological or psychiatric disease
* American Society of Anaesthesiologists (ASA) classification greater than or equal to class IV
* Moribund patients

Due to the underlying PKPD models of the SmartPilot® system, patient with the following characteristics cannot be anesthetized using SmartPilot®:

* Height < 150 or > 200 cm, respectively
* Weight < 40 or > 140 kg, respectively
* Body Mass Index > 30
* Age < 18 or > 90 years of age, respectively

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male/female patients scheduled for elective surgery (general/abdominal surgery; traumatological/orthopedic surgery, gynecology, urology) in general anesthesia at Charité - Universitaetsmedizin Berlin, Campus Mitte and Campus Virchow-Klinikum
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2013-11-12 (Actual); Primary Completion 2016-03-01 (Actual); Study Completion 2017-07-14 (Actual)

PRIMARY OUTCOMES:
Postoperative delirium | In the 8-day postoperative sample period
  Nursing Delirium Csreening Scale (Nu-DESC), Confusion Assessment Method for the Intensive Care Unit (CAM-ICU), Diagnostic and Statistical Manual of Mental Disorders (DSM-IV-R), International Classification of Diseases (ICD-10)
Postoperative cognitive deficit | In the 8-day postoperative sample period
  Test Battery: Verbal Learning Test, Stroop Colour Word Test, Letter Digit Substitution Test, Concept Shifting Test

SECONDARY OUTCOMES:
Wake-up time | In the 8-day postoperative sample period
Duration of treatment in the recovery room | In the 8-day postoperative sample period
Correlation of EEG-based depth of anesthesia (BIS®) with PK/PD-based Noxious Stimulus Response Index (NSRI) of the SmartPilot® system. | In the 8-day postoperative sample period
Correlation of Bispectral index (BIS®)- and NSRI readings with Near infrared spectroscopy (NIRS) - readings as parameters of regional cerebral oxygen saturation. | In the 8-day postoperative sample period

CONTACTS AND LOCATIONS:
Overall Officials: Spies Claudia, MD, Prof., Study Director — Charite University, Berlin, Germany
Locations (1):
- Department of Anesthesiology and Intensive Care Medicine, Campus Virchow Klinikum, Charité - Universitätsmedizin, Berlin, Germany